CLINICAL TRIAL: NCT06740266
Title: The Impact of Stress and Caregiver Sensitivity on Infant Cellular Aging in a Population of Under-Resourced Families: A Randomized Controlled Trial
Brief Title: The Impact of an Evidence-Based Parenting Service on Maternal Sensitivity and Infant Cellular Aging in a Population of Under-Resourced Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: WakeMed Health and Hospitals (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Monica Oxford, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00019057; R01NR021020 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Parent Child Relationship; Child Social-Emotional Development; Telomere Length; Epigenetic Aging
Keywords: Epigenetic aging; Parenting intervention; Parent sensitivity; Pediatric setting
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promoting First Relationships in Primary Care (PFR-PC) (Experimental): PFR is a strengths-based, evidence-based home visiting approach to engage with families in ways that promote positive parenting change. PFR is a manualized training curriculum consisting of a 10-week (1 hour per visit) intervention. Each week has a theme for discussion and an activity. During five of the weekly sessions, the provider videotapes playtime between mother and child. On alternate weeks, the PFR provider and the mother watch the videotaped playtime and reflect about the needs of both the mother and the child. PFR-PC adds two additional visits at the medical home during routine well-child visits. PFR-PC is a manualized primary care delivery model with content that corresponds to developmentally appropriate content aligned with the well-child visits. Each family will receive two sessions at WakeMed during their well-child visits (approximately 20 minutes in length).
  Interventions: Behavioral: Promoting First Relationships in Primary Care (PFR-PC)
- Usual care (No Intervention): Usual care consists of routine pediatric medical well and sick care from WakeMed pediatrics, as well as already existing onsite integrated mental health and social work services.

INTERVENTIONS:
Behavioral: Promoting First Relationships in Primary Care (PFR-PC) — Promoting First Relationships® in Primary Care is based on attachment theory and is strengths-based. The intervention is delivered in 10 home visits, with 2 additional clinic visits. Each week has a theme for discussion, handouts, an activity, and time for "joining" - checking in with the parent, listening to their concerns, and establishing a positive, supportive relationship. The provider videotapes playtime between parent and child, and alternates weeks watching the video with the parent, reflecting about the needs of both parent and child (reflective observation). PFR consultation strategies include Joining, Positive Feedback, Instructive Feedback, Reflective Questions and Comments, and Instruction with Handouts. These core strategies enhance parents' sense of security and competency. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent to identify their own feelings and needs around parenting.
  Arms: Promoting First Relationships in Primary Care (PFR-PC)

SUMMARY:
The goal of this clinical trial study is to learn how stress in childhood, or Early Life Adversity (ELA), gets "under the skin" and influences long-term health. The investigators will test if the support given to parents of young children reduces childhood stress. The investigators will also test if the effects of mother's stress and Early Life Adversity can be passed down to children. Can it impact the child's long-term health? Researchers will compare the Promoting First Relationships® in Primary Care (PFR in PC) parenting program with Usual Care to see if PFR reduces mothers' stress, improves mother's sensitivity, and reduces accelerated cellular aging.

Participants will:

* Be randomized to receive PFR in PC or Usual Care. PFR in PC is an evidence-based 10-week home visiting service, with 2 extra sessions at the WakeMed pediatric clinic. Usual Care is the health care and general services offered to families at the WakeMed pediatric clinic.
* Have in-home research visits at the start of the study (Time 1, T1), about 6 months later (Time 2, T2), and 12 months later (Time 3, T3). Information collected at these visits includes:

  * Answering questions about your background, past and current stress, physical and mental health, parenting behaviors, and child behavior problems (T1, T2, T3).
  * Being videotaped doing a short teaching activity.
  * Having a small amount of blood collected from the mother by finger prick (T1, T3).
  * Having a small amount of blood collected from the infant by heel stick (T1, T3).

DETAILED DESCRIPTION:
Early life adversity (ELA) is a salient risk factor for later-life morbidity and early mortality. During the first years of life, children are particularly vulnerable to adverse events. Notably, these adversities are disproportionately placed on families of color and can lead to health disparities. Cellular aging is a potential mechanism by which ELA confers lifelong risks. Interventions implemented during sensitive developmental periods early in life may yield a higher efficacy and reduce health disparities. The aim of the proposed randomized controlled trial (RCT) is to test if an evidence-based home visiting model, Promoting First Relationships® (PFR), that improves caregiver sensitive and responsive care, when embedded within a primary care setting, will protect young infants from the effect of stress on accelerated cellular aging.

Telomeres, the structures at the end of chromosomes, are considered a marker for cellular aging. Telomeres shorten with each cell division and this can lead to cellular senescence, one of the key hallmarks of aging. Shorter telomere length (TL) is associated with poorer physical and mental health outcomes. In addition to TL, "epigenetic clocks", which are composed of dozens or hundreds of methylation marks, predict mortality and are linked with disability and disease processes. There is preliminary evidence that epigenetic age (EpiAge) is accelerated by perinatal risk exposures and lifetime adversity, and that stress-related mechanisms forecast accelerated EpiAge. The literature has shown that TL and EpiAge are malleable and receptive to environmental inputs, interventions that focus on family support and a healthy lifestyle, as well as parental sensitivity, which operates as a protective factor.

The investigators have an incredible opportunity to advance the field to understand the impact of past and present stressors, caregiver sensitive and responsive care, on infant cellular aging (including both TL and EpiAge clocks), in a sample of under-resourced families receiving PFR through their primary care setting. PFR is a 10-week home visiting model that has, in five prior RCTs, consistently improved caregiver sensitivity and responsive care, as well as parental knowledge of children's social-emotional needs. PFR has shown improvements at the biological level in children through Respiratory Sinus Arrhythmia, a marker of emotional regulation, and stimulated cortisol responses. This study will expand upon these findings and will be the first to evaluate PFR, delivered in the context of primary care (PFR-PC), on children's cellular aging.

The setting for this study is unique. WakeMed Primary Care in North Carolina is a busy pediatric practice that utilizes an integrated care model to serve a high-need patient population. Their aim is to reduce disparities through services embedded within primary care. WakeMed's pediatric practice serves nearly 7,000 families in one of the highest-need zip codes in the state. Of their highly diverse patients, 90% receive Medicaid. Embedding PFR within a primary care setting is an innovative strategy to facilitate an integrated care model and to enhance resilency in minoritized lower income families. In this RCT, we will recruit a low-income, community sample of 250 Spanish- and English-Speaking mothers and their infants receiving primary care from WakeMed. Mothers will be randomized to Usual Care (UC) or to PFR in Primary Care (PFR-PC) 10-week home visiting with follow-up content during two well-child visits. We will collect dried blood spots from mothers and children to evaluate TL and various EpiAge clocks. We will also advance the literature by accounting for important heritability factors (i.e., maternal TL at baseline) and intergenerational controls (i.e., maternal Adverse Childhood Experiences (ACEs) and paternal age at conception). The investigators will measure mothers' TL at baseline and child TL and EpiAge clocks at baseline and one-year post-baseline.

Aim 1: Evaluate three under-studied heritability and intergenerational predictors of cellular aging: Test whether 1) maternal TL, 2) maternal ACEs, and 3) paternal age at conception predict child baseline TL. It is hypothesize that heritability and intergenerational measures will predict child baseline TL. The investigators will further evaluate the effect of maternal ACEs on child EpiAge clocks at baseline.

Aim 2: Evaluate the impact of adversity on change in cellular aging. We will test if current adversity (caregiver depression, discrimination, violence, and difficult life events) predicts child cellular aging (TL and EpiAge clocks) between baseline and 12 months post-enrollment, controlling for heritability and intergenerational effects (Aim 1) and PFR-PC. It is hypothesize that children exposed to greater concurrent adversity will evidence accelerated cellular aging compared with children with less adversity.

Aim 3: Test whether PFR-PC reduces accelerated cellular aging. Test PFR-PC on change in TL and EpiAge among children in a population with high health disparities one-year post-intervention. It is hypothesize that 1) children in the PFR-PC treatment group will have significantly longer TL and younger EpiAge than those in the UC control group 1-year post enrollment. It is also hypothesize that 2) treatment difference in TL/EpiAge will be mediated by maternal sensitivity using standard mediation and that PFR will improve mother sensitivity and child behavior. Exploratory aim. Evaluate PFR-PC implementation (dosage, quality, acceptability, satisfaction, and provider fidelity). Based on prior studies, it is hypothesize that PFR will demonstrate successful implementation (dosage, quality, acceptability, satisfaction, and provider fidelity).

ELIGIBILITY:
Inclusion Criteria:

* Biological mother of infant aged 3-12 months English- or Spanish-speaking Receiving Medicaid Their infant is receiving pediatric care at WakeMed

Exclusion Criteria:

* Experiencing an acute crisis (e.g. hospitalization, incarceration) Homeless or without stable enough housing for home visits Lacking access to a phone Previously received the Promoting First Relationships intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Telomere length change | Baseline (Time 1), 12-months post-baseline (Time 3)
  DNA will be extracted from DBS samples using Qiagen's QIAamp DNA Mini Kit. Extracted DNA is quantified using a NanoDrop 2000 spectrophotometer (Thermo Fisher), checked for integrity using TapeStation bioanalyzer and Quant-iT Picogreen (Invitrogen) to specifically determine double-stranded DNA concentration.
EpiAge clock change | Baseline (Time 1), 12-months post-baseline (Time 3)
  DNAm will be determined using the Illumina Infinium Methylation EPIC v2.0 BeadChip Array (llumina Inc, CA) at Pennsylvania State University's genomics core lab. Arrays are processed using the Illumina iScan platform according to the manufacturer's protocol.
Maternal sensitive and responsive care change | Baseline (Time 1), 6- months post baseline (Time 2), 12-months post-baseline (Time 3)
  Parent sensitivity is measured by the Nursing Child Assessment Teaching Scale (NCATS; Barnard 1994), a videotaped interaction to assess caregiver sensitivity, stimulation of the child, and emotional responsiveness during interaction. The range of this scale is zero to 73, higher scores indicate greater sensitivity
Maternal Knowledge of Social and Emotional Development change | Baseline (Time 1), 6- months post baseline (Time 2), 12-months post-baseline (Time 3)
  16-item Likert-scale questionnaire developed by the study, "Raising a Baby." The scale is summed, and scores could range from 16 to 64, with higher scores indicating greater parental knowledge.

SECONDARY OUTCOMES:
Child Behavior Problems change | Baseline (Time 1), 6- months post baseline (Time 2), 12-months post-baseline (Time 3)
  The Infant-Toddler Social and Emotional Assessment (ITSEA) in English or Spanish is a standard child assessment tool assessing emotional and behavioral problems in young children. The ITSEA has been standardized and normed on a nationally representative sample that was stratified to match the 2002 U.S. Census. Mothers rated their infant on an extensive list of behaviors from 0 (not true/rarely) to 2 (very true/often). T scores are calculated. Higher T scores indicate more problem behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Oxford, PhD, Principal Investigator — University of Washington
Locations (1):
- WakeMed Health & Hospitals, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are looking into the mechanisms and details for doing this, in consultation with the University and in accordance with NIH policies. We will update this section when this has been worked out.